CLINICAL TRIAL: NCT03830307
Title: An Open-Label Application of the NSS-Bridge Device for Post-Cesarean Pain
Brief Title: NSS-Bridge Device for Post-Cesarean Delivery Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grace Lim, MD, MS (Other)
Responsible Party: Sponsor-Investigator, Grace Lim, MD, MS, Director of Obstetric Anesthesia, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19010299
Record Dates: First submitted 2019-02-01; First posted 2019-02-05 (Actual); Results first posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Acute Pain; Cesarean Delivery
Keywords: Pain Therapy; Auriculotherapy; Cesarean Delivery
MeSH Terms: conditions — Acute Pain; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Intervention Group (Experimental): The NSS-2 BRIDGE is a battery operated and disposable percutaneous auricular nerve field stimulator (Innovative Health Solutions, Versailles, IN, USA), that was recently cleared by the FDA and assigned a Class II Risk Designation; a class which includes surgical drapes, pumps and power wheelchairs. The indication for the NSS-2 BRIDGE is for the treatment of clinical symptoms related to opioid consumption and opioid withdrawal.
  Interventions: Device: NSS-2-Bridge

INTERVENTIONS:
Device: NSS-2-Bridge — NSS-2-Bridge auricular therapy will be given in addition to standard of care

SUMMARY:
The current opioid epidemic has led to a renewed interest in exploring non-pharmacological techniques to treat post-operative pain. An increasing number of patients are suffering from the adverse effects of opioid use following surgery, including post-operative nausea and vomiting, respiratory depression, immunosuppression, constipation, and most recently, addiction. In the United States, over $600 billion is spent every year on opioid addiction, including $79 billion related to opioid addiction following surgery. Despite many initiatives to decrease the use of opiates in the preoperative setting, opioids continue to be regularly prescribed before, during and after surgery. Although the risk of opioid addiction following surgery is recognized, the percentage of patients becoming addicted to opioids following surgery is not well understood. To date, there has been virtually no agreement regarding the duration and dosage that qualify for opioid dependence following surgery, nor that a clear estimation of the factors such as biological, psychosocial and socioeconomic that increase the risk of using opioids for extended periods of time after surgery. Therefore, in order to combat this growing health crisis at the ground level, it is incumbent upon the medical community to explore alternative methods of pain control to treat the surgical population in order to reduce the incidence of post-operative opioid addiction.

Percutaneous Nerve Field Stimulation (PNFS) is one of these recognized methods that ongoing research has shown to be effective as a complementary method of pain management. While PNFS is not a novel concept, clinical indications of auricular field stimulation have been limited in the past due to requirement of bulky, stationary and non-disposable stimulators and electrodes. These technological limitations made it difficult to establish the real clinical potential of auricular stimulation for the perioperative management of pain in surgical patients, despite the demonstration that auriculotherapy has been shown to relieve pain in the postoperative setting.

The NSS-2 BRIDGE is a battery operated and disposable percutaneous auricular nerve field stimulator (Innovative Health Solutions, Versailles, IN, USA), that was recently cleared by the FDA and assigned a Class II Risk Designation; a class which includes surgical drapes, pumps and power wheelchairs. The indication for the NSS-2 BRIDGE is for the treatment of clinical symptoms related to opioid consumption and opioid withdrawal. These symptoms include abdominal pain, anxiety and post-operative nausea and vomiting; conditions which are also present following cesarean-section surgery. The use of the NSS-2 BRIDGE device has been demonstrated to provide significant analgesia in patients with abdominal pain syndrome, and clinical trials are ongoing to assess the benefit of this approach for post-operative pain management. As compared to the present use of opioids for perioperative pain management, the use of a complementary, non-pharmacologic approach offers the advantage of analgesia without the associated side effects.

DETAILED DESCRIPTION:
The primary purpose of this pilot study is to demonstrate feasibility/acceptability of the BRIDGE device as applied after cesarean delivery. Once the feasibility/acceptability is confirmed, the cesarean delivery model will be included in an NIH application related to the use of devices to reduce opioid use. In this pilot period, no changes will be made in the other routine analgesia/postpartum care. Following the same previously published approaches from our group, potential subjects will be recruited in the Magee-Womens Hospital obstetrical unit when they arrive for cesarean delivery. Patients will be asked if they are interested in using the BRIDGE system as a way to control pain after the cesarean delivery. They will be offered the option to review a video explaining the mechanism of action if the BRIDGE system. They will also be provided with information about the acceptability of the BRIDGE device in other clinical settings. Subjects will be informed of the purpose of this pilot evaluation and signed written informed consent to participate in the study.

Once the subject has given and signed informed consent to participate in the study, demographic information and medical history will be collected from each participant on the day of the cesarean delivery. Data will be de-identified and kept in a locked cabinet and secured servers. The NSS-2 BRIDGE device will be applied to one ear by trained research staff in the immediate post-operative setting. The patient will be informed at the time of consent and after the implantation of the device that they can have the device removed anytime after its application.

Per current standard of care, pain will be assessed in the postpartum period. At 24, 48, 72, 96 and 120 hours post-operatively the investigators will collected pain scores at rest and movement, pain unpleasantness, total opioid consumption (from the medical record), as well as the devise tolerability.

The investigators will also collect common medical information including time to bowel movement, postoperative nausea and vomiting (PONV), time to oral intake (liquid and regular diet), time to hospital discharge, overall patient satisfaction, and patient satisfaction related to pain management. When the patient is discharged from the hospital, they will be asked to complete a patient satisfaction survey. For patients discharged with the device attached, removal instructions will be given to patient to remove and dispose of the device at 120 hours.

Standard opioid conversion table will be used to convert the oral and IV narcotic utilized by the patients to IV morphine equivalent doses (MED) for analysis purposes.

Overall patient satisfaction and satisfaction of pain management during hospitalization will be measured by a numerical rating scale with 0 being worst satisfaction and 10 being the best satisfaction. The patient satisfaction test will be administered by a member of the research team.

No statistical analysis will be performed. The primary end point for this pilot phase will be the descriptive feasibility and acceptability of the use of this device un cesarean delivery population. We will assess the experience of device tolerability along with pain intensity. Pain intensity scores and opioid consumption will be compared to data obtained from historical data of women undergoing cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Cesarean delivery

Exclusion Criteria:

* History of active depression, anxiety or catastrophizing
* Active alcoholism or drug abuse
* Severe chronic pain condition that requires daily preoperative opioid use
* Current opioid maintenance therapy/use for any other reason
* History of hemophilia
* Patients with cardiac pacemakers
* Patients with psoriasis vulgaris diagnosis or other skin conditions affecting the ear

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2019-04-04 (Actual); Study Completion 2019-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace Lim, MD, MS, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period was from 3/11/2019-3/29/2019
Period: Overall Study
Arm/Group | Intervention Group
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Group
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption
Description: Investigate the efficacy of the NSS-2 BRIDGE device in reducing perioperative opioid consumption in opioid-naïve patients undergoing elective cesarean section surgery using the current post-operative standard of care.
Time Frame: Day of surgery through post-operative day 5
Measure: Mean (Full Range); unit: milligrams of oxycodone
Arm/Group | Intervention Group
Number analyzed (Participants) | 5
milligrams of oxycodone | 31 [0 to 60]

2. Secondary Outcome: Number of Participants With Post-operative Complications
Description: Investigate the incidence of post-operative complications for patients receiving the NSS-2-Bridge device.
Time Frame: Day of Surgery through 90 days post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 5
Participants | 0

3. Secondary Outcome: Efficacy of NSS-2 Bridge Device: Opioid Consumption
Description: Investigate the efficacy of the NSS-2 BRIDGE device in changing perioperative opioid consumption in opioid-naïve patients undergoing elective cesarean section surgery.
Time Frame: Day of Surgery through 90 days post-operative
Population: 90 follow-up of opioid medication was not collected in intervention group
Arm/Group | Intervention Group
Number analyzed (Participants) | 0

4. Secondary Outcome: Level of Comfort Wearing NSS-2 Bridge Device
Description: Level of comfort while wearing device will be evaluated by a score on a scale (0- no discomfort 10- worst discomfort). The minimum value is 0 and the maximum value is 10. Higher scores mean a worse outcome.
Time Frame: 24 hours post-operatively
Population: Some participants were unavailable to give a discomfort score on some days, hence the discrepancy of the number analyzed versus overall enrolled
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 4
score on a scale | 1.5 [0 to 4]

5. Secondary Outcome: Level of Comfort Wearing NSS-2 Bridge Device
Description: as for outcome 4
Time Frame: 48 hours post-operatively
Population: as for outcome 4
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 3
score on a scale | 0 [0 to 8]

6. Secondary Outcome: Level of Comfort Wearing NSS-2 Bridge Device
Description: as for outcome 4
Time Frame: 72 hours post-operatively
Population: as for outcome 4
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 3
score on a scale | 0 [0 to 0]

7. Secondary Outcome: Level of Comfort Wearing NSS-2 Bridge Device
Description: as for outcome 4
Time Frame: 96 hours post-operatively
Population: as for outcome 4
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 2
score on a scale | 1 [0 to 2]

8. Secondary Outcome: Level of Comfort Wearing NSS-2 Bridge Device
Description: as for outcome 4
Time Frame: 120 hours post-operatively
Population: as for outcome 4
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 3
score on a scale | 0 [0 to 0]

9. Secondary Outcome: Pain Score at Rest
Description: Pain Score at rest will be measured by a score on a scale (0=no pain 10=most pain). The minimum value is 0 and the maximum value is 10. Higher scores mean a worse outcome.
Time Frame: 24 hours post-operatively
Population: Some participants were unavailable to give a pain score on some days, hence the discrepancy of the number analyzed versus overall enrolled
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 5
score on a scale | 0 [0 to 7]

10. Secondary Outcome: Pain Score at Rest
Description: as for outcome 9
Time Frame: 48 hours post-operatively
Population: as for outcome 9
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 5
score on a scale | 4 [2 to 8]

11. Secondary Outcome: Pain Score at Rest
Description: as for outcome 9
Time Frame: 72 hours post-operatively
Population: as for outcome 9
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 4
score on a scale | 3 [0 to 4]

12. Secondary Outcome: Pain Score at Rest
Description: as for outcome 9
Time Frame: 96 hours post-operatively
Population: as for outcome 9
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 2
score on a scale | 1 [0 to 2]

13. Secondary Outcome: Pain Score at Rest
Description: =Pain Score at rest will be measured by a score on a scale (0=no pain 10=most pain). The minimum value is 0 and the maximum value is 10. Higher scores mean a worse outcome.
Time Frame: 120 hours post-operatively
Population: as for outcome 9
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 3
score on a scale | 0 [0 to 2]

14. Secondary Outcome: Pain Score With Movement
Description: Pain Score with movement will be measured by a score on a scale (0=no pain 10=most pain). The minimum value is 0 and the maximum value is 10. Higher scores mean a worse outcome.
Time Frame: 24 hours post-operatively
Population: as for outcome 9
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 4
score on a scale | 4 [0 to 7]

15. Secondary Outcome: Pain Score With Movement
Description: as for outcome 14
Time Frame: 48 hours post-operatively
Population: as for outcome 9
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 3
score on a scale | 4 [2 to 10]

16. Secondary Outcome: Pain Score With Movement
Description: as for outcome 14
Time Frame: 72 hours post-operatively
Population: as for outcome 9
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 3
score on a scale | 5 [2 to 7]

17. Secondary Outcome: Pain Score With Movement
Description: as for outcome 14
Time Frame: 96 hours post-operatively
Population: as for outcome 9
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 2
score on a scale | 2.5 [2 to 3]

18. Secondary Outcome: Pain Score With Movement
Description: as for outcome 14
Time Frame: 120 hours post-operatively
Population: as for outcome 9
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 3
score on a scale | 2 [2 to 3]

ADVERSE EVENTS:
Time Frame: 90 days
Description: The subjects' medical record charts were reviewed daily by research staff and any findings would be assessed by the principal investigator.
Arm/Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT03830307/Prot_000.pdf